CLINICAL TRIAL: NCT01009099
Title: Reducing Dynamic Hyperinflation Through Breathing Retraining
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F6955-R
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Pulmonary Disease; COPD
Keywords: pulmonary disease; COPD
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): exercise training with breathing retraining
  Interventions: Other: breathing retraining; Other: exercise training
- Arm 2 (Active Comparator): exercise training
  Interventions: Other: exercise training

INTERVENTIONS:
Other: breathing retraining — breathing retraining using a metronome
  Arms: Arm 1
Other: exercise training — treadmill exercise training

SUMMARY:
This study will compare the effects of exercise training and breathing retraining (using metronome tones) to exercise training only. Exercise training lasts 12 weeks.

DETAILED DESCRIPTION:
Dynamic hyperinflation limits exercise tolerance in chronic obstructive pulmonary disease (COPD). To limit dynamic hyperinflation during exercise and thus improve exercise tolerance, we successfully developed a visual-auditory ventilation-feedback system. The system retrains patient's breathing pattern during exercise. The goal of the current proposal was to develop a user-friendly ventilation-feedback technique with a novel auditory feedback system. We reasoned that the proposed feedback system plus exercise training would be superior to exercise training alone while having the potential for an easier application into clinical practice. Hypotheses: The primary hypothesis is that the exercise duration of patients with moderate-to-severe COPD who successfully complete a 12-week program of breathing retraining plus exercise will be longer than that of patients who complete a 12-week program of treadmill exercise training alone. We also hypothesized that the primary predictor of improved exercise duration will be a reduction in dynamic hyperinflation and to a lesser extent, improvement in peripheral muscle function. Lastly, we hypothesize that dyspnea will be reduced in patients assigned to breathing retraining plus exercise when compared to exercise training alone. Methods: The proposed study was a randomized controlled clinical trial. 119 patients with moderate-to-severe COPD were randomized into breathing retraining plus exercise or exercise training alone. Both groups received 12-weeks of treadmill exercise training three times weekly. The breathing retraining plus exercise group also received auditory feedback to decrease respiratory rate and prolong exhalation. The goal of breathing retraining was to reduce exercise-induced dynamic hyperinflation. Follow-up testing was completed at 6, 12, and 24 weeks. Testing included a pulmonary function test, symptom-limited and constant workrate treadmill tests, six-minute walk, dyspnea measurements, testing of respiratory muscle strength and endurance, and quadriceps muscle endurance testing. Analysis: Measures of central tendency will be used to describe the study sample. A two-sample t-test ( = 0.05) was used to analyze changes from baseline to 12-weeks between the breathing retraining plus exercise group and exercise training alone group. In data analysis, intention-to-treat principles were used. Since several measures will be taken on each patient, mixed-models analysis will be used to compare changes over time between the two groups. Multiple regression analysis will be employed to determine the predictors of improved exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* 40 yr of age
* FEV1 70%
* FEV1/FVC < 70%
* RV/TLC 120%
* mean SpO2 90% at peak exercise (w/ or w/o O2)
* Able to hear metronome sounds Lives near Hines, IL (Chicagoland area)

Exclusion Criteria:

* Respiratory infection/exacerbation within the previous four weeks
* Exercise limiting heart disease (+ stress test or other indicators of heart disease or complaints of angina during the stress test)
* Primary asthma
* Congestive heart failure (New York Heart Association Class III or IV)
* Exercise-limiting peripheral arterial disease (stops exercise due to intermittent claudication)
* Stops exercise due to arthritic pain in the knee or hips (self-report)
* Inability to walk on the treadmill
* Pregnancy
* Any unforeseen illness or disability that would preclude exercise testing or training
* Participation in a formal exercise program within the previous 12 weeks

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen G. Collins, PhD RN, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

REFERENCES:
- [Derived] Collins EG, Jelinek C, O'Connell S, Butler J, Reda D, Laghi F. The Effect of Breathing Retraining Using Metronome-Based Acoustic Feedback on Exercise Endurance in COPD: A Randomized Trial. Lung. 2019 Apr;197(2):181-188. doi: 10.1007/s00408-019-00198-4. Epub 2019 Feb 9. PMID 30739217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from a midwestern VA hospital and were also referred from other patients and private practices.
Pre-assignment Details: 204 patients signed informed consents and were screened for participation in the study. 85 patients did not meet eligibility criteria for the following reasons: PFT results did not meet study criteria, claudication, cardiac issues, non-compliance, changed their mind, and active substance use. 119 patients were enrolled in the protocol.
Groups:
- Exercise Training With Breathing Retraining: treadmill exercise training plus breathing retraining using a metranome
Period: Overall Study
Arm/Group | Exercise Training With Breathing Retraining | Exercise Training
Started | 58 | 61
Completed | 53 | 57
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 58 | 61 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.9) | 66.3 (8.1) | 66.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 54 | 59 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 57 | 61 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 14 | 30
  White | 42 | 47 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 61 | 119
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.0 (6.7) | 29.3 (6.2) | 29.7 (6.5)
FEV1 [Mean (Standard Deviation); unit: percent predicted] | 43.7 (14.9) | 44.0 (13.9) | 43.8 (14.3)
FEV1/FVC [Mean (Standard Deviation); unit: percent] | 46.6 (13.3) | 45.1 (12.1) | 45.8 (12.7)
RV/TLC [Mean (Standard Deviation); unit: percent predicted] | 171.3 (30.3) | 168.2 (26.6) | 169.7 (28.4)
Peak oxygen uptake [Mean (Standard Deviation); unit: VO2 mL/kg/min] | 15.7 (3.9) | 16.6 (3.3) | 16.1 (3.6)
Time on treadmill constant workrate test [Mean (Standard Deviation); unit: minutes walked] | 6.8 (2.5) | 6.9 (2.3) | 6.9 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Exercise Duration (Time Walked on the Constant Workrate Treadmill Test)
Description: The primary outcome measure is a comparison of time walked on the constant workrate treadmill best at 12 weeks.
Time Frame: baseline and 12 weeks
Population: Patients who completed 12 weeks of exercise training were analyzed. There was one patient in each group that did not complete the treadmill test at 12 weeks although they completed other secondary outcome measures. Although they did not complete this measure, they remained in the study and were not counted as a drop.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Exercise Training With Breathing Retraining | Exercise Training
Number analyzed (Participants) | 52 | 56
minutes | 15.2 (14.8) | 17.6 (14.1)
Statistical Analysis 1: Comparison: Exercise Training With Breathing Retraining vs Exercise Training; The outcomes compared were time walked on the constant workrate treadmill test measured in minutes; Test type: Superiority or Other; p = 0.63, ANCOVA; Co-variates included in the analysis were time walked on the constant workrate test at baseline and adherence (sessions completed/expected)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 6 months (baseline through end of study or 6 months).
Arm/Group | Exercise Training With Breathing Retraining | Exercise Training
Serious Adverse Events (participants affected / at risk) | 1/58 | 5/61
Other Adverse Events (participants affected / at risk) | 2/58 | 5/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise Training With Breathing Retraining (N=58) | Exercise Training (N=61)
ischemic cerebrovascular (Nervous system disorders) | 0 | 2 — Transischemic attack (TIA)
fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 — Fractured rib (fall on ice)
pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — patient went to ED for muscle soreness
arterial injury-extremity lower (Vascular disorders) | 0 | 1 — Iliac artery aneurysm identified
infection peripheral nerve (Infections and infestations) | 0 | 1 — herpes zoster
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Training With Breathing Retraining (N=58) | Exercise Training (N=61)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes